CLINICAL TRIAL: NCT02307955
Title: Firefly ANKLE Sprain Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKD-ffANK-001
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Grade I/II Ankle Sprain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- firefly (Experimental): participants treated with firefly device
  Interventions: Device: firefly
- Control (Other): Standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: firefly
  Arms: firefly
Other: Standard of care
  Arms: Control

SUMMARY:
The device to be tested (fireflyTM) stimulates the common peroneal nerve and causes the foot to twitch, and has been shown to increase blood flow. The device is also indicated for the treatment of oedema. In this study the investigators intend to assess the use of the device as an adjunctive therapy for people recovering from grade 1 and 2 ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. Referred to physiotherapy for treatment of ankle sprain
3. Clinical diagnosed ankle sprain with evidence of swelling
4. Able to understand the Subject Information Sheet and willing to sign the written Informed Consent Form.
5. Able and willing to follow the protocol requirements

Exclusion Criteria:

1. Has an ankle sprain grade 3
2. Evidence of fracture
3. Has a pacemaker
4. Chronic Obesity (BMI Index >40kg/m2).
5. Pregnancy.
6. History or signs of previous deep or superficial vein thrombosis/pulmonary embolism.
7. Varicosities, ulceration or erosion around the area of the leg where the study device would be fitted
8. Not able to fit firefly device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Oedema lower leg | 1 week
FAAM ankle function measure | 1 week

SECONDARY OUTCOMES:
Ankle proprioception - as assessed by the time that the participant can stand on one leg for with their eyes closed, this will be recorded and repeated three times, the average will be taken | 1 week
VAS Pain score | 1 week
Adverse event rate | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Poole NHS Trust Hospital, Poole, Dorset, United Kingdom